CLINICAL TRIAL: NCT05040737
Title: Comparison of Two Types of Dialyzers (PMMA vs Polysulfone) on Cytokine Extraction in Hemodialysis Patients and COVID Infection. A Multicenter Prospective Study
Brief Title: PMMA vs Polysulfone in SARS-CoV-2 Infection Hemodialysis Patients
Acronym: Dial-COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Mª Jesús Puchades, MD PhD, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Dial-COVID
Record Dates: First submitted 2021-08-01; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: SARS-CoV-2 Infection
Keywords: Haemodialysis; SARS-CoV-2 Infection; cytokines
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Patients will be dialysed according to the usual dialysis schedule of three weekly sessions. The study has a duration of 8 days in order to include 4 haemodialysis sessions. The first and third haemodialysis sessions will be dialysed with PS membrane and the second and fourth sessions with PMMA membrane, both dialysers with a surface area of 1.8 m2.
  Interventions: Device: PS membrane versus PMMA membrane,

INTERVENTIONS:
Device: PS membrane versus PMMA membrane, — Patients will be dialysed according to the usual dialysis schedule of three weekly sessions. The study has a duration of 8 days in order to include 4 haemodialysis sessions. The first and third haemodialysis sessions will be dialysed with PS membrane and the second and fourth sessions with PMMA membrane, both dialysers with a surface area of 1.8 m2.

SUMMARY:
Controlled, prospective, open-label trial with a total duration of 2 weeks to assess the clearance of inflammatory interleukins by different membranes in haemodialysis patients with COVID-19.

DETAILED DESCRIPTION:
Controlled, prospective, open-label trial with a total duration of 2 weeks to assess the clearance of inflammatory interleukins by different membranes in haemodialysis patients with COVID-19.

Patients will be dialysed according to the usual dialysis schedule of three weekly sessions. The study has a duration of 8 days in order to include 4 haemodialysis sessions. The first and third haemodialysis sessions will be dialysed with PS membrane and the second and fourth sessions with PMMA membrane, both dialysers with a surface area of 1.8 m2.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years .
* Patient on chronic haemodialysis admitted to the hospital with a diagnosis of infection by COVID-19.
* Signature of informed consent or legal representative.
* Estimated duration of admission greater than 8 days (4 haemodialysis sessions).
* Patient with haemodynamic stability, understood as systolic blood pressure ≥ 100 mmHg.

Exclusion Criteria:

* Refusal to sign the consent form.
* Patients who for clinical reasons are unable to follow a regular dialysis schedule of three sessions per week.
* Allergy (documented or suspected) to either of the two membranes involved in the study.
* Patient with haemodynamic instability (Mean arterial pressure < 100 mmHg).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Inflammatory interleukins reduction with two different dialysis membranes (PMMA and PS). | Day 8
  To compare the percentage reduction of inflammatory interleukins measured at the beginning and end of haemodialysis in the same patient with COVID 19 infection dialysed with two different dialysis membranes (PMMA and PS).

SECONDARY OUTCOMES:
Percentage of Inflammatory interleukins reduction | Days 5 and 8
  Inflammatory interleukins reduction maintenance with each membrane after a second dialysis
Inflammatory interleukins reduction (30 minutes) | Days 1,3,5,8
  Inflammatory interleukins percentage reduction 30 min after each session,
Populational characteristics | Day 8
  To describe the characteristics of haemodialysis population affected by COVID -19

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Valencia, Spain